CLINICAL TRIAL: NCT03262246
Title: Cerebral Infarction and White Substance in Angiopathy Cerebral Amyloid
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ISAAC
Record Dates: First submitted 2017-08-24; First posted 2017-08-25 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-08

CONDITIONS: Amyloid Angiopathy
MeSH Terms: conditions — Amyloid angiopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: medical report consultation — investigators consult medical report concerning patient identified for cerebral amyloid angiopathy

SUMMARY:
The cerebral amyloïd angiopathy ( AAC) is a disease characterized by deposits of beta-amyloid peptids in the walls of the arteries of young and average calibre of the brain and the leptomeninx. The incidence of the AAC increases strongly with the age and represents a major cause of spontaneous brain haemorrhage to people over 60. The main demonstration is the lobar brain haemorrhage, the other ones are bleedings under arachnoid cortical and microbleedings leading to cognitive decline.

Anatomical studies reported the presence of cortical infarcts in patients having amyloïd deposits suggesting an association between asymptomatic cortical cerebral infarcts and AAC.

However prevalence and meaning of these infarcts in patients having an AAC remain badly known because of studies on low number of patients and the rarity of radiological analyses of these infarcts .A better knowledge of these asymptomatic cortical infarcts would allow to dread better cognitive disorders(confusions) presented by these patients, and to develop preventive strategies.

Besides, the risk factors of severity of the AAC are little studied.

ELIGIBILITY:
Inclusion Criteria:

* age>55
* hospitalized in CAEN hospital and Paris St Joseph Hospital between 1st january 2011 and 31 december 2015 for cerebral haemorrhage with MRI images diagnosing cerebral amyloid angiopathy.

Exclusion Criteria:

* Insufficient MRI images quality without FLAI sequence, T2 GRE
* disease with same radiologic and clinical signs that cerebral amyloid angiopathy.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators select medical report of hospitalized patient between 2011/01/01 and 2015/12/31 in CAEN hospital and Paris St Joseph hospital ; these had an MRI for cerebral haemorrhage.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
number of patient with cerebral infarction and associated factors in a cohort of cerebral amyloid angiopathy patients | 1day

CONTACTS AND LOCATIONS:
Overall Officials: HODEL Jérome, Professor, Principal Investigator — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France